CLINICAL TRIAL: NCT03646149
Title: Improving Housing Outcomes for Homeless Veterans (CDA 15-074)
Brief Title: Improving Housing Outcomes for Homeless Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 18-004; CDA 15-074 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-04

CONDITIONS: Veterans; Homeless Persons; Mentally Ill Persons
Keywords: Social Skills; Housing
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Housing Skills Training Group Patients (Experimental): Homeless Veterans with serious mental illness who are inpatient at the VA Greater Los Angeles Domiciliary or enrolled in a VA Supported Housing (VASH) program and participating in a Housing Skills Training Group as part of routine clinical care. The intervention was 12 sessions long, with one session per week.
  Interventions: Behavioral: Housing Skills Training Group

INTERVENTIONS:
Behavioral: Housing Skills Training Group — 12-session social skills training group for persons with homeless experiences and serious mental illness delivered once a week for 12 weeks

SUMMARY:
Many homeless Veterans with serious mental illness (SMI) enroll in the VA's Supported Housing (VASH) program but struggle to obtain and sustain housing. Social skills are an important-but underappreciated-determinant of housing outcomes for homeless adults. The investigators hypothesize that homeless Veterans with SMI who participate in a social skills training program, tailored for housing-related social skills, will obtain housing quicker, retain housing longer, and show improved mental health outcomes compared to Veterans with similar needs not participating in such a program.

ELIGIBILITY:
Inclusion Criteria:

* Identified by VA Greater Los Angeles homeless program staff as a participant in Housing Skills Training:

  * Must have a history of homelessness
  * Must be a Veteran over the age of 18 years
  * Must have a serious mental illness (mood disorder, anxiety disorder, psychotic disorder)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Emi Gabrielian, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will create de-identified, study-specific datasets that include all variables in a publication. Some loss of information might occur given the need to remove PHI. The PI will replace social security and medical station numbers with study-specific numbers. The PI will drop date of birth and replace age with age categories, in accordance with PHI requirements for people 85 years of age and older. Dates of service will be replaced with year dummies.
Time Frame: Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication.
Access Criteria: Prior to distribution, a local privacy officer will certify that all datasets contains no PHI. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Letter of Agreement.

REFERENCES:
- [Derived] Gabrielian S, Hamilton AB, Gelberg L, Koosis ER, Hoffmann L, Carlson DM, Young AS. Testing an implementation package in a housing skills training pilot for homeless-experienced persons with serious mental illness. Implement Res Pract. 2024 Mar 6;5:26334895241236679. doi: 10.1177/26334895241236679. eCollection 2024 Jan-Dec. PMID 38449910

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Providers were not enrolled in the study. The investigators collected outcome data about perceived impressions / satisfaction with the intervention, from providers, but did not collect any information about their baseline characteristics (these were providers who provided this intervention as part of routine clinical care in an implementation pilot but who were not engaged in research) and do not consider them an arm in this intervention or those outcomes to be part of this clinical trial
Groups:
- Housing Skills Training Group: Homeless Veterans with serious mental illness who are inpatient at the VA Greater Los Angeles Domiciliary or enrolled in a VA Supported Housing (VASH) program and participating in a Housing Skills Training Group as part of routine clinical care.
Period: Overall Study
Arm/Group | Housing Skills Training Group
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline data collection was only performed on the Veteran (patient) group. The providers were engaged in data collection post-intervention but not baseline data collection
Groups:
- Housing Skills Training Patients: Homeless Veterans with serious mental illness who are inpatient at the VA Greater Los Angeles Domiciliary or enrolled in a VA Supported Housing (VASH) program and participating in a Housing Skills Training Group as part of routine clinical care. Though providers completed one outcome variable for this study to report on their satisfaction with the intervention (an early implementation outcome) they were not considered a distinct arm in this trial.
Arm/Group | Housing Skills Training Patients
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity : Hispanic or Latino | 2
  Ethnicity : Not Hispanic or Latino | 32
  Ethnicity : Decline to state | 1
  Race: African American | 24
  Race: White | 10
  Race: Multiracial | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35
Percent service-connected disability [Count of Participants; unit: Participants]
  0% | 11
  10-30% | 3
  40-60% | 6
  70-100% | 15
Current housing status [Count of Participants; unit: Participants]
  Stable housing | 7
  Sheltered housing | 27
  Unsheltered homeless | 1
Mental health diagnoses [Number; unit: participants]
  Depression | 21
  Bipolar disorders | 1
  Post-traumatic stress disorder | 20
  Anxiety disorders | 4
  Schizophrenia and other psychotic disorders | 4
Substance use disorders [Number; unit: participants]
  Drug use disorders | 27
  Alcohol use disorders | 19

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire - 8
Description: Acceptability of the intervention to participants Scores range from 8 to 32, with higher values indicating higher satisfaction (no specific cut-offs to indicate specific levels of satisfaction)
Time Frame: 12 weeks after baseline assessment at start of intervention
Population: Only 16 patients agreed to fill out this voluntary outcome measure at the completion of the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Housing Skills Training Patients: Homeless Veterans with serious mental illness who are inpatient at the VA Greater Los Angeles Domiciliary or enrolled in a VA Supported Housing (VASH) program and participating in a Housing Skills Training Group as part of routine clinical care.
Arm/Group | Housing Skills Training Patients
Number analyzed (Participants) | 16
score on a scale | 26.2 (4.1)

2. Secondary Outcome: Percent Days Housed for One Year After Intervention Completion
Description: We will use the medical record, augmented by the residential time line follow back, to assess longitudinal housing outcomes for Veterans receiving this intervention
Time Frame: 1 year
Population: Due to the COVID-19 pandemic, we were unable to engage in face-to-face interaction with participants to obtain 1-year post intervention housing data
Arm/Group | Housing Skills Training Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Housing Skills Training Group
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03646149/Prot_SAP_000.pdf